CLINICAL TRIAL: NCT00001041
Title: Active Immunization of HIV-1 Infected, Pregnant Women With CD4 Lymphocyte Counts >= 400/mm3: A Phase I Study of Safety and Immunogenicity of MN rgp120/HIV-1 Vaccine (NOTE: Some Patients Receive Placebo)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Model: Parallel | Purpose: Prevention
Other Study IDs: ACTG 235; AVEG 104; 11212 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Pregnancy
Keywords: Vaccines, Synthetic; Pregnancy; Pregnancy Complications, Infectious; HIV Envelope Protein gp120; AIDS Vaccines; HIV Therapeutic Vaccine
MeSH Terms: conditions — HIV Infections; Pregnancy Complications, Infectious

INTERVENTIONS:
Biological: rgp120/HIV-1MN

SUMMARY:
To evaluate the safety of rgp120/HIV-1MN vaccine in HIV-1 infected pregnant women with CD4 counts >= 400 cells/mm3. To evaluate the immunogenicity of this vaccine in pregnant women and the passive acquisition of vaccine-specific antibody in their infants. To evaluate the induction or augmentation by rgp120/HIV-1MN vaccine of mucosal immune response in the gastrointestinal and reproductive tracts during pregnancy. To isolate and genetically characterize the HIV-1 present in cervicovaginal fluid specimens of pregnant women and compare it to that present in their peripheral blood mononuclear cells and to that of their infected infants.

Evidence suggests that an advanced stage of disease with high plasma viremia is associated with increased transmission of HIV-1 to the fetus. Slowing the progression of disease, reducing the titer of virus in plasma, and increasing the titer of epitope-specific antibody are potentially attainable goals through active immunization of the mother during pregnancy.

DETAILED DESCRIPTION:
Evidence suggests that an advanced stage of disease with high plasma viremia is associated with increased transmission of HIV-1 to the fetus. Slowing the progression of disease, reducing the titer of virus in plasma, and increasing the titer of epitope-specific antibody are potentially attainable goals through active immunization of the mother during pregnancy.

Pregnant women are randomized to receive an initial injection of MN rgp120 vaccine or alum placebo between week 16 and week 24 of gestation, followed by monthly booster injections concluding at the end of pregnancy, for a total of five injections. Patients may have optional booster immunizations (vaccine or placebo) at 3, 6, 9, and 12 months after delivery. Mothers and infants are followed through 18 months after delivery. Per 06/94 addendum, patients will be contacted once or twice per year for at least 5 years to check on health status of patient and child. PER 12/21/94 ADDENDUM, post-partum immunizations are discontinued.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* AZT.
* Acyclovir.

Patients must have:

* HIV-1 infection.
* CD4 count >= 400 cells/mm3.
* No AIDS-defining illness or other systemic manifestations related to HIV (other than generalized lymphadenopathy).
* HIV p24 < 30 pg/ml.
* Proven pregnancy in the 16th to 24th week of gestation at study entry, with no special obstetrical risks.
* Concurrent AZT therapy is permitted.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms and conditions are excluded:

* Known hypersensitivity to a component of the vaccine.
* Evidence of fetal abnormality on ultrasound.
* Evidence of maternal risk factors including insulin-dependent diabetes, moderate to severe hypertension, repeated fetal wastage (> 3), Rh-sensitization or other blood group alloimmunization, severe renal disease, previous infants with malformations or other factors that obstetrically are judged to constitute a special risk of spontaneous abortion or premature birth.
* Active syphilis.
* Hepatitis B surface antigen positive.

Concurrent Medication:

Excluded:

* Antiretroviral or immunomodulating agent other than AZT during the pregnancy.

Prior Medication:

Excluded:

* Antiretroviral or immunomodulating agent other than AZT within 90 days prior to study entry.

Current use of illicit drugs or known chronic alcohol use.

Ages: 16 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24
Dates: Study Completion 1998-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wara DW, Study Chair; Lambert JS, Study Chair; Wright PF, Study Chair
Locations (6):
- United States (6):
  - San Francisco Gen. Hosp., San Francisco, California
  - UCSF Pediatric AIDS CRS, San Francisco, California
  - Johns Hopkins Hosp. & Health System - Dept. of Peds., Div. of Infectious Diseases, Baltimore, Maryland
  - Washington U CRS, St Louis, Missouri
  - St. Louis ConnectCare, Infectious Diseases Clinic, St Louis, Missouri
  - Univ. of Rochester ACTG CRS, Rochester, New York

REFERENCES:
- [Derived] Hompe ED, Mangold JF, Kumar A, Eudailey JA, McGuire E, Haynes BF, Moody MA, Wright PF, Fouda GG, Giorgi EE, Gao F, Permar SR. Induction of Neutralizing Responses against Autologous Virus in Maternal HIV Vaccine Trials. mSphere. 2020 Jun 3;5(3):e00254-20. doi: 10.1128/mSphere.00254-20. PMID 32493720